CLINICAL TRIAL: NCT02139124
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Multi-Center Study Measuring the Efficacy and Safety of PRC-063 in Adult ADHD Patients
Brief Title: The Efficacy and Safety of PRC-063 in Adult ADHD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Collaborators: Purdue Pharma, Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 063-010
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo
- PRC-063 25 mg (Experimental): PRC-063 25 mg
  Interventions: Drug: PRC-063 25 mg
- PRC-063 45 mg (Active Comparator): PRC-063 45 mg
  Interventions: Drug: PRC-063 45 mg
- PRC-063 70 mg (Active Comparator): PRC-063 70 mg
  Interventions: Drug: PRC-063 70 mg
- PRC-063 100 mg (Active Comparator): PRC-063 100 mg
  Interventions: Drug: PRC-063 100 mg

INTERVENTIONS:
Drug: Placebo — Oral placebo capsule
  Other Names: Placebo capsule
  Arms: Placebo
Drug: PRC-063 25 mg — Oral 25 mg capsule - active
  Other Names: 25 mg capsule
  Arms: PRC-063 25 mg
Drug: PRC-063 45 mg — Oral 45 mg capsule - active
  Other Names: 45 mg capsule
  Arms: PRC-063 45 mg
Drug: PRC-063 70 mg — Oral 70 mg capsule - active
  Other Names: 70 mg capsule
  Arms: PRC-063 70 mg
Drug: PRC-063 100 mg — Oral 100 mg capsule - active
  Other Names: 100 mg capsule
  Arms: PRC-063 100 mg

SUMMARY:
The purpose of this randomized, placebo-controlled, double-blind, parallel group study is to evaluate the clinical efficacy and safety of PRC-063 in adults with ADHD

DETAILED DESCRIPTION:
This study is a randomized, phase III, multicenter, placebo-controlled, parallel-group, forced-dose titration in which adult subjects (18 years of age or older) with ADHD will be randomized to PRC-063 (25, 45, 70 or 100 mg) or placebo for four weeks of double-blind evaluation of safety and efficacy. The study will have four phases: (1) screening and 1-week washout; (2)baseline and double-blind, forced-dose titration over a 2-week period; (3) double-blind evaluation over a 2-week period; and (4) a 14-day safety follow-up. Subjects will be required to visit the site 6 times over a 5 week period.

Screening and Washout: Subjects will be screened to establish eligibility for study participation. Subjects who meet eligibility requirements will undergo ADHD medication washout, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female at least 18 years of age and meeting the local, legal definition of adult.
* ADHD diagnosis, inattentive, hyperactive/impulsive or combined, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) based on clinician assessment using multiple informants and a structured interview.
* Unsatisfied with his or her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects naïve to pharmacological therapy for ADHD is permitted.
* Female subjects must be one of the following: a. surgically sterile prior to screening; b.

postmenopausal; c. if of childbearing potential, abstinent or willing to use a reliable method of contraception, such as oral contraceptive, two barrier methods, a barrier method plus a spermicidal agent.

* Female subjects of Child-Bearing Potential (FOCP) must have a negative serum β-hCG pregnancy test at screening.
* Minimum level of intellectual functioning, as determined by an Intelligence Quotient (IQ) score of 80 or above based on the WASI.
* Mentally and physically competent to sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Able and willing to comply with the study procedures for the entire length of the study, including a successful swallow test of an empty 100 mg capsule.

Exclusion Criteria:

* Having an allergy to methylphenidate or amphetamines or a history of serious adverse reactions to methylphenidate.
* Known to be non-responsive to methylphenidate treatment. Non-response is defined as methylphenidate use at various doses for a phase of at least four weeks at each dose with little or no clinical benefit.
* Being diagnosed with or having a history of strokes, epilepsy, migraine headaches (greater than 1 instance every two months), glaucoma, thyrotoxicosis, tachyarrhythmias or severe angina pectoris or serious or unstable medical illness. Subjects with controlled or stable asthma or diabetes will be permitted.
* Elevated blood pressure, defined as any values above 89 diastolic or 139 systolic, as assessed at Visit 1.
* Clinically significant ECG abnormalities, as assessed at Visit 1.
* Clinically significant laboratory abnormalities, as assessed at Visit 1.
* Currently receiving guanethidine, pressor agents, MAO inhibitors, coumarin anticoagulants, anticonvulsants (e.g. phenobarbital, phenytoin, primidone), phenylbutazone, tricyclic antidepressants (e.g. imipramine, desipramine), selective serotonin reuptake inhibitors (SSRIs) or herbal remedies (unless on a stable dose for 4 weeks).
* Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary heart disease, transient ischemic attack or stroke or other serious cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subjects who are currently considered a suicide risk by the investigator.
* Having a primary diagnosis of schizophrenia, schizoaffective disorder, primary affective disorder, schizotypal personality, major depression, bipolar disorder, generalized anxiety, borderline personality disorder, antisocial personality or another unstable psychiatric condition requiring treatment, as assessed by the structured interview conducted at Visit 1.
* Having a history or suspected physiological dependence (excluding nicotine) on narcotic analgesics or other psychoactive drugs (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines).
* Excessive consumption of alcohol (consumes alcohol in quantities greater than 15 drinks per week; 1 drink is defined as 360 mL/12 oz. of beer, 120 mL/4 oz. of wine, or 30 mL/1 oz. of hard liquor), or history (within previous 6 months) of alcohol abuse.
* Currently (or within 30 days before the planned start of treatment) receiving an investigational drug or using an experimental medical device.
* Homeless.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Reiz, Study Director — Purdue Pharma LP
Locations (38):
- United States (33):
  - UCLA, Los Angeles, California
  - Synergy Clinical Research, National City, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Orange County Neuro Phychiatry Research Centre, Orange, California
  - Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Research, Gainesville, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - CNS Healthcare Jacksonville, Jacksonville, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Advanced Clinical Research, Boise, Idaho
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Princeton Medical Institute, Princeton, New Jersey
  - Medical Research Network, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigation, Portland, Oregon
  - Oregon Center for Clinical Investigation, Salem, Oregon
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Bayou City Research Ltd, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Houston Clinical Trials, Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Ericksen Research, Clinton, Utah
  - Physiciatric and Behavioral Solutions, Salt Lake City, Utah
  - Woodstock Research Center at Neuropsychiatric Associates, Woodstock, Vermont
  - NeuroScience, Herndon, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
- Canada (5):
  - Dr. Margaret Weiss, Vancouver, British Columbia
  - Doctors Jackiewicz Professional Medical Corporation, Niagara Falls, Ontario
  - Dr. Judy van Stralen, Ottawa, Ontario
  - The Kids Clinic, Whitby, Ontario
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss MD, Surman C, Khullar A, He E, Cataldo M, Donnelly G. Effect of a Multi-Layer, Extended-Release Methylphenidate Formulation (PRC-063) on Sleep in Adults with ADHD: A Randomized, Double-Blind, Forced-Dose, Placebo-Controlled Trial Followed by a 6-month Open-Label Extension. CNS Drugs. 2021 Jun;35(6):667-679. doi: 10.1007/s40263-021-00814-z. Epub 2021 May 31. PMID 34057707

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | PRC-063 25 mg | PRC-063 45 mg | PRC-063 70 mg | PRC-063 100 mg
Started | 78 | 77 | 73 | 73 | 74
Completed | 69 | 73 | 69 | 61 | 61
Not Completed | 9 | 4 | 4 | 12 | 13
Not completed — Adverse Event | 2 | 0 | 1 | 2 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1
Not completed — non-compliant | 1 | 0 | 0 | 2 | 0
Not completed — incarceration | 0 | 0 | 1 | 0 | 0
Not completed — subject moved | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PRC-063 25 mg | PRC-063 45 mg | PRC-063 70 mg | PRC-063 100 mg | Total
Number analyzed (Participants) | 78 | 77 | 73 | 73 | 74 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.4) | 36.3 (12.48) | 36.0 (11.82) | 35.1 (11.19) | 35.3 (11.68) | 36.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 36 | 35 | 44 | 198
  Male | 35 | 37 | 37 | 38 | 30 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 6 | 13 | 14 | 52
  Not Hispanic or Latino | 68 | 66 | 66 | 60 | 58 | 318
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 3 | 0 | 2 | 3 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 9 | 8 | 13 | 1 | 10 | 41
  White | 64 | 69 | 57 | 68 | 59 | 317
  More than one race | 1 | 0 | 1 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-administered ADHD-5-Rating Scale Total Score
Description: Participants were monitored for 4 weeks on treatment (final 2 weeks on stable dose). Clinicians rated subject behavior on the ADHD-5-Rating Scale each week. Primary outcome was based on the final week of treatment. The ADHD-5-RS is an 18-item questionnaire that measures the frequency of ADHD symptoms based on DSM-5 criteria. For each item, clinicians rate how often the behavior is displayed on a scale of 0 (Never or Rarely) to 3 (Very Often). Scores can range from 0 to 54, with lower scores indicating a lower frequency of ADHD symptoms.
Time Frame: 4 weeks
Population: The Full Analysis population consists of all randomized subjects who receive any amount of study medication and who have any ADHD-5-Rating Scale assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 0 mg/Day: Placebo
Arm/Group | PRC-063 25 mg | PRC-063 45 mg | PRC-063 70 mg | PRC-063 100 mg | 0 mg/Day
Number analyzed (Participants) | 77 | 73 | 73 | 74 | 78
units on a scale | 24.2 (11.88) | 19.9 (12.45) | 24.0 (11.25) | 18.7 (11.48) | 26.1 (11.99)
Statistical Analysis 1: Comparison: PRC-063 25 mg vs 0 mg/Day; The null hypothesis is "the mean Clinician ADHD-5-RS total score at Visit 6 is not different between the active treatment and placebo."; Test type: Superiority; p = 0.6750, ANCOVA — The model includes terms for treatment and baseline Clinician ADHD-5-RS score as a covariate; Analyses utilize ANCOVA models with Dunnett's adjustments for multiple pairwise comparisons for each active dose group with placebo; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-6.6 to 2.6]
Statistical Analysis 2: Comparison: PRC-063 45 mg vs 0 mg/Day; The null hypothesis is the mean Clinician ADHD-5-RS total score at Visit 6 is not different between the active treatment and placebo; Test type: Superiority; p = 0.0013, ANCOVA — The model includes terms for treatment and baseline Clinician ADHD-5-RS score as a covariate; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-11.5 to -2.2]
Statistical Analysis 3: Comparison: PRC-063 70 mg vs 0 mg/Day; The null hypothesis is "the mean Clinician ADHD-5-RS total score at Visit 6 is not different between the active treatment and placebo"; Test type: Superiority; p = 0.6720, ANCOVA — The model includes terms for treatment and baseline Clinician ADHD-5-RS score as a covariate; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-6.8 to 2.7]
Statistical Analysis 4: Comparison: PRC-063 100 mg vs 0 mg/Day; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0002, ANCOVA — The model include terms for treatment and baseline Clinician ADHD-5-RS score as a covariate; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-12.9 to -3.2]

ADVERSE EVENTS:
Time Frame: double blind phase
Arm/Group | Placebo | PRC-063 25 mg | PRC-063 45 mg | PRC-063 70 mg | PRC-063 100 mg
Serious Adverse Events (participants affected / at risk) | 2/78 | 4/77 | 2/73 | 2/73 | 4/74
Other Adverse Events (participants affected / at risk) | 25/78 | 30/77 | 36/73 | 45/73 | 47/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | PRC-063 25 mg (N=77) | PRC-063 45 mg (N=73) | PRC-063 70 mg (N=73) | PRC-063 100 mg (N=74)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | PRC-063 25 mg (N=77) | PRC-063 45 mg (N=73) | PRC-063 70 mg (N=73) | PRC-063 100 mg (N=74)
conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (3)
dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (5) | 5 (5) | 9 (9)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (5) | 2 (2) | 8 (9)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
energy increased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 6 (6)
feeling jittery (General disorders) | 1 (1) | 1 (1) | 1 (1) | 6 (7) | 3 (3)
pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
alanine aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blood creatine phosphokinase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
blood pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
heart rate increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
weight decreased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 5 (5) | 11 (11) | 14 (14)
increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
disturbance in attention (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 8 (9) | 7 (8) | 14 (18) | 15 (15) | 9 (9)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mental impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
restless leg syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
bruxism (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
initial insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 6 (6) | 4 (4) | 5 (6)
insomnia (Psychiatric disorders) | 2 (2) | 12 (12) | 8 (9) | 11 (12) | 14 (16)
irritability (Psychiatric disorders) | 3 (3) | 7 (7) | 5 (5) | 2 (3) | 2 (2)
middle insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
orgasm abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No